CLINICAL TRIAL: NCT00852111
Title: Molecular-Genetic Correlates of Fatigue in Cancer Patients Receiving Localized External Beam Radiation Therapy
Status: Completed | Type: Observational
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090088; 09-NR-0088
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Fatigue
Keywords: Fatigue; Radiotherapy; Cancer Therapy; Natural History; Cancer
MeSH Terms: conditions — Neoplasms; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Prostate cancer patients

SUMMARY:
Background:

* Researchers have studied the causes of fatigue during treatments for various diseases, but these results have not been conclusive.
* More information on the physical changes that affect the body during treatment may help identify biological or chemical factors that contribute to patient fatigue, which may allow physicians to identify individuals who may be more at risk of feeling fatigue before, during, and after treatment for diseases such as cancer.

Objectives:

* To identify factors contributing to fatigue in men who are undergoing radiation treatment for prostate cancer.

Eligibility:

* Men 18 years of age and older who are scheduled to receive localized radiation treatment for prostate cancer.

Design:

* Six outpatient visits to the NIH Clinical Center, approximately on the same day and same time of day:
* First visit before beginning radiation treatment.
* Once a week for the first 2 weeks of the treatment, once at the midpoint of treatment, once at the end of treatment.
* Final visit 4 weeks after completion of radiation treatment.
* Initial visit will involve a physical examination and questions about medical history.
* Evaluations during the treatment period:
* Blood draws to identify cells and chemicals associated with inflammation and fatigue.
* Questions about physical activity, fatigue, depression, and quality of life.

DETAILED DESCRIPTION:
Although the underlying mechanisms of fatigue have been studied in several disease conditions the data are not conclusive, and this symptom remains poorly managed at present. Longitudinal studies related to treatment-related fatigue in prostate cancer patients have been conducted, but there are limited studies exploring the changes in physiologic mechanisms before and after radiotherapy which can identify individuals who are at risk for enduring fatigue during and after therapy. Fatigue is conceptualized as a multidimensional symptom which incorporates temporal, sensory, cognitive/mental, affective/emotional, behavioral, and physiological dimensions. This prospective, observational study is the first study to explore the molecular-genetic mechanisms underlying fatigue and the cluster of symptoms (urinary, sexual, gastrointestinal, psychiatric) experienced by prostate cancer patients undergoing External Beam Radiation Therapy (EBRT).

The primary objective of the study is to describe the changes in the self-reported fatigue; urinary, sexual, and gastrointestinal symptoms; depression; fatigue catastrophizing; and health-related quality of life (HRQOL) experienced by patients with and without prostate surgery before, during, and after EBRT completion. The secondary objectives of this study are to investigate the pro-inflammatory cytokine profile of EBRT-related fatigue (TNF alpha, IGF-I, IL-6, IL-8, TGF alpha and beta), determine changes in white blood cell gene expression, determine levels of oxidative stress and changes in potential biomarkers influencing oxidative stress from blood and buccal samples before and after EBRT completion and to relate these changes in the levels of these biological markers to self-reported fatigue; urinary, sexual, and gastrointestinal symptoms; depression; fatigue catastrophizing; and HRQOL scores. This study also aims to measure the skeletal muscle strength, activity/fitness levels, cognitive function and energy expenditure of patients before, at completion of EBRT, and at least 6 months post EBRT and relate these findings with self-reported fatigue, physical symptoms (e.g. urinary, gastrointestinal, and sexual functioning), depression, and HRQOL scores before and after an exercise training program. The study also aims to describe changes in chemical profile in the brain that are associated with changes in fatigue symptoms using magnetic resonance spectroscopy before and after EBRT.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be included, patients must meet all of the following criteria:

* Clinically localized prostate cancer with or without prior prostatectomy;
* Scheduled to receive EBRT either by 3D conformal or IMRT techniques that is not anticipated to change during the course of the study, with or without ADT;
* No known medical history of tuberculosis (TB);
* Able to provide written informed consent by passing at least 80% of the consent quiz;
* Greater than or equal to18 years of age;

The control group must meet all the inclusion criteria mentioned above except for number 2. The control group must not be receiving any form of treatment for their prostate cancer to include hormone, immune, radiation, or chemotherapy.

EXCLUSION CRITERIA:

All participants with any one of the following criteria will be excluded:

Progressive or unstable disease of any body system causing clinically significant fatigue, including cardiovascular, pulmonary, gastrointestinal, central nervous system, psychiatric, endocrine, hematologic, renal, or immunologic disorders, and including patients with any of the following broad disease categories:

* Systemic infections (e.g., human immunodeficiency virus (HIV), active hepatitis);
* Documented history of major depression, bipolar disease, psychosis, or alcohol dependence/abuse within the past 5 years;
* Uncorrected hypothyroidism and anemia;
* Chronic inflammatory disease that may be anticipated to alter the proinflammatory cytokine profile (i.e. rheumatoid arthritis, systemic lupus erythematosus, and cirrhosis).

Patients taking tranquilizers, steroids, and nonsteroidal anti-inflammatory agents because these medications are known to affect cytokine production;

Patients who have second malignancies or those receiving chemotherapy with their EBRT.

In addition to the above criteria, participants with the following conditions will be excluded from participating in the exercise interventions:

1. Significant Restrictive or Obstructive Lung Disease
2. Ischemic heart disease
3. Left ventricular dysfunction
4. Acute corpulmonale
5. Cardiomyopathy (dilated, hypertrophic, or non-idiopathic)
6. Significant renal or hepatic dysfunction
7. Disabling stroke
8. Uncontrolled diabetes mellitus with a history of diabetic ketoacidosis
9. Mitochondrial disease

Participants unable to pass the English comprehension test will be unable to take the Computer Assessment of Mild Cognitive Impairement (CAMCT) test but will be asked to complete the other outcome measures of the study.

Self report of color-blindness, verified by taking the Ishihara card test and scoring greater than 14 (more or less than 10 minutes), will exclude a participant from taking the STROOP test, but will be asked to complete the other outcome measures of the study. This card test will be administered only if the patient states they are color blind.

- Individuals capable of becoming pregnant.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This protocol will enroll 262 men with prostate cancer, 161 (116 without prior prostatectomy and 45 with previous prostatectomy) who are scheduled to receive EBRT. Additional 56 men will be invited to participate in 8-week, an hour/day, 3 days/week aerobic exercise programs (CT [N=28], HIIT [N=28]). It will also enroll 45 men with prostate cancer who are not currently receiving any treatment to serve as the control group for the study. Ten additional prostate cancer subjects (with and without previous prostatectomy) who are scheduled to be treated with EBRT will also be enrolled for the pilot study subgroup to determine associations between fatigue with structural and chemical changes of the brain using magnetic resonance spectrospcopy (MRS). Thirty additional men (with and without previous prostatectomy) will be enrolled for the pilot study subgroup to collect buccal swabs to measure proteins related to mitochondrial function. The study will enroll a total of 262 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2009-04-23 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Change in Fatigue Score measured by PROMIS-Fatigue scale | Ongoing

SECONDARY OUTCOMES:
Change in gene expression, cytokine profile, skeletal muscle strength, cognitive function | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Leorey N Saligan, C.R.N.P., Principal Investigator — National Institute of Nursing Research (NINR)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-NR-0088.html